CLINICAL TRIAL: NCT00013858
Title: Environmental Contaminants and Infant Development
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Indian and Northern Affairs, Canada (Other); Health Canada (Other Government); Danish Institute for Public Health (Other)
Other Study IDs: 7902-CP-001
Record Dates: First submitted 2001-03-30; First posted 2001-04-03 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Mercury Poisoning; Lead Poisoning
Keywords: methylmercury; PCBs; lead; fish consumption; breast-feeding
MeSH Terms: conditions — Mercury Poisoning; Lead Poisoning; Breast Feeding

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is designed to examine the effects of prenatal exposure to environmental contaminants on cognitive and behavioral development and physical growth in two groups of Inuit infants-one in Northern Quebec; the other in Greenland.

DETAILED DESCRIPTION:
Due to prevailing weather patterns and ocean currents, certain environmental contaminants are transported to the Arctic region. The Inuit are among the most heavily exposed populations on earth due to the prevalence of these contaminants in traditional foods that comprise a large portion of their diet. The contaminants assessed in this study include polychlorinated biphenyls (PCBs), methylmercury, selenium, organochlorine pesticides, and lead. These contaminants are measured in umbilical cord blood samples obtained at birth, milk samples obtained from breast-feeding mothers and, in the case of mercury, hair samples obtained from the mothers. Omega-3 and omega-6 fatty acids are also assessed in these samples to examine the degree to which these nutrients may protect against adverse effects attributable to these contaminants.

ELIGIBILITY:
infant born during recruitment period to a mother who is a resident of Povungnituk, Inukjuak, and Kuujjuarapik, Quebec or Nuuk, Greenland

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 1997-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Centre of Quebec, Beauport, Quebec, Canada

REFERENCES:
- [Background] Dewailly, E., Bruneau, S., Ayotte, P., Liliberte, C., Gingras, S. Belander, D. and Ferron, L. Health status at birth of Inuit newborn prenatally exposed to organochlorines - Chemosphre, 1993, 27: 359-366.
- [Background] Dewailly E, Ayotte P, Bruneau S, Laliberte C, Muir DC, Norstrom RJ. Inuit exposure to organochlorines through the aquatic food chain in arctic quebec. Environ Health Perspect. 1993 Dec;101(7):618-20. doi: 10.1289/ehp.93101618. PMID 8143594
- [Background] Jacobson SW, Fein GG, Jacobson JL, Schwartz PM, Dowler JK. The effect of intrauterine PCB exposure on visual recognition memory. Child Dev. 1985 Aug;56(4):853-60. PMID 3930167
- [Background] Jacobson JL, Jacobson SW. Intellectual impairment in children exposed to polychlorinated biphenyls in utero. N Engl J Med. 1996 Sep 12;335(11):783-9. doi: 10.1056/NEJM199609123351104. PMID 8703183